CLINICAL TRIAL: NCT06913829
Title: Efficacy Of Pencil Pushup Exercise Vs Base Out Exercising Prism's In Patient With Convergence Insufficiency
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/811
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Convergence Insufficiency
MeSH Terms: conditions — Ocular Motility Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- base-out exercising prisms (Experimental)
  Interventions: Combination Product: base-out exercising prisms
- pencil pushup exercises (Active Comparator)
  Interventions: Diagnostic Test: pencil pushup exercises

INTERVENTIONS:
Combination Product: base-out exercising prisms — Participants in the experimental group will use base-out exercising prisms as their primary intervention. This involves:
  1. Procedure:
     * Wearing customized prism glasses designed to increase the convergence demand during near tasks.
     * Performing near vision activities such as reading or viewing objects while wearing the prisms.
  2. Schedule:
     * Prisms will be prescribed based on individual clinical measurements.
     * Participants will use the prisms during near tasks for 15-20 minutes daily, 5 days a week, for a total duration of 6 weeks.
  3. Monitoring:
     * Initial training will be provided to ensure proper use of the prisms.
     * Adherence will be checked during weekly follow-up visits, where adjustments to the prism strength will be made if necessary.
  Arms: base-out exercising prisms
Diagnostic Test: pencil pushup exercises — Participants in the control group will perform pencil pushup exercises as their primary intervention. This involves: 1. Procedure: o Holding a pencil or similar object vertically at arm's length and focusing on a letter or small mark on it. o Gradually moving the pencil closer to the nose until the participant experiences visual blur or sees double. o Returning the pencil to the starting position and repeating the process. 2. Schedule: o Exercises will be prescribed for 15-20 minutes daily, 5 days a week, for a total duration of 6 weeks. 3. Monitoring: o Participants will receive instructions during the initial session and periodic supervision at follow-up visits to ensure proper technique and adherence. o Progress will be monitored weekly through symptom reporting and clinical measurements.
  Arms: pencil pushup exercises

SUMMARY:
Convergence insufficiency (CI) is a prevalent binocular vision disorder that leads to symptoms such as eye strain, headaches, and blurred vision during near work. This study aims to evaluate and compare the efficacy of pencil pushup exercises versus base-out exercising prisms in the management of CI. A Randomized Controlled Trial (RCT) will be conducted with 28 participants, using non-probability convenience sampling from SIGHTON Optix, Lahore. Participants will be randomly assigned to either the experimental group (receiving base-out exercising prisms) or the control group (receiving pencil push up exercises). The study will assess symptom improvement using the Convergence Insufficiency Symptom Survey (CISS), near point of convergence (NPC).

DETAILED DESCRIPTION:
The study will also evaluate quality of life (QoL) using a vision-related QoL questionnaire. The total study duration is 3 months, with a primary goal of determining the relative efficacy of these two interventions. This study is expected to provide valuable insights into effective, evidence-based management options for convergence insufficiency, ultimately improving patient outcomes and guiding clinical practice. The collected data will be analysed by using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Patients having CISS score more than 16 or higher for children aged <21 and 21 or higher for adults.
* Patients diagnosed with convergence insufficiency based on clinical tests (e.g., near point of convergence).
* Age group: 10-50
* Patients experiencing symptoms related to convergence insufficiency, such as eye strain, headaches, blurred vision, or double vision during near work.
* Able to perform pencil push-up exercises correctly after demonstration.
* No other significant ocular or neurological conditions that might affect vision or convergence.

Exclusion Criteria:

* Any type of strabismus.
* Amblyopia.
* Refractive error more than 6 diopters.
* Patients with history of prism prescription.
* History of strabismus surgery or refractive error surgery.
* History of eye trauma.
* Any systemic and neurological diseases affecting binocular vision such as diabetes, myasthenia gravis, Graves', and multiple sclerosis.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Convergence Insufficiency Symptom Survey | 12 Months
  For Children (< age 21) total score = 16 or higher is suggestive of convergence insufficiency. For Adults total score = 21 or higher is suggestive of convergence insufficiency.
Quality of Life Questionnaire (QOL) | 12 Months
  Scoring Instructions:
  * Each response is scored on a scale from 1 to 5, based on the patient's answer.
  * A higher score indicates a greater negative impact on quality of life.
  Interpretation:
  * Low Scores (10-20): Minimal impact on quality of life.
  * Moderate Scores (21-35): Moderate impact on daily life and well-being.
  * High Scores (36-50): Significant impact on daily activities and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- SIGHTON Optix Mozang Chungi, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No